CLINICAL TRIAL: NCT00231283
Title: A Multicenter, Non-Randomized Study of the CYPHER NxT Sirolimus-Eluting Coronary Stent on BX SONIC OVER-THE-WIRE (OTW) Stent Delivery System(SDS)for the Treatment of de Novo Native Coronary Artery Lesions
Brief Title: NEXUS Study for the Treatment of de Novo Native Coronary Artery Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sidney Cohen, MD, PhD, Vice President, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04-6324
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2010-03-23 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): CYPHER NxT Sirolimus-eluting Coronary Stent on the BX SONIC Over-the-wire Stent Delivery System
  Interventions: Device: CYPHER NxT SES ON BX SONIC OTW STENT DELIVERY SYSTEM (SDS)

INTERVENTIONS:
Device: CYPHER NxT SES ON BX SONIC OTW STENT DELIVERY SYSTEM (SDS) — CYPHER NxT Sirolimus-eluting Coronary Stent on the BX SONIC Over-the-wire Stent Delivery System

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of the CYPHER NxT Sirolimus-eluting Coronary Stent on the BX SONIC Over-the-Wire (OTW) Stent Delivery System (SDS) in patients with de novo native coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female patients 18 years of age
2. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;
3. Treatment of a single de novo target lesion in a major native coronary artery;
4. Target lesion is 2.5 mm and 3.5 mm in diameter (visual estimate);
5. Target lesion is 30mm in length (visual estimate);
6. Target lesion stenosis is > 50% and < 100% (visual estimate);

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK > 2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remain above normal at the time of treatment;
2. Has unstable angina classified as Braunwald III B or C, or is having a peri-infarction angina;
3. Significant (> 50%) stenoses proximal or distal to the target lesion that might require revascularization or impede runoff;
4. Documented Left ventricular ejection fraction 25%;
5. Totally occluded vessel (TIMI 0 level);
6. Impaired renal function (creatinine > 3.0 mg/dl) at the time of treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-04; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD, Principal Investigator — Texas Heart Institute
Locations (1):
- Texas Heart Institute, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled was Apr 2004 and last patient enrolled was Jul 2004.
Groups:
- CYPHER NxT Stent on the BX SONIC OTW SDS: CYPHER NxT Sirolimus-eluting Coronary Stent on the BX SONIC Over-the-wire Stent Delivery System
Period: Overall Study
Arm/Group | CYPHER NxT Stent on the BX SONIC OTW SDS
Started | 100
Completed | 95
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | CYPHER NxT Stent on the BX SONIC OTW SDS
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 64.39 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 68
Region of Enrollment [Number; unit: participants]
  United States | 100
Patients with Diabetes Mellitus [Number; unit: participants]
  With Diabetes Mellitus | 25
  Without Diabetes Mellitus | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Procedure Success From Post-procedure to Hospital Discharge
Description: Procedure Success is defined as the final residual diameter stenosis < 50 percent by Quantitative Coronary Angiography (QCA) using any percutaneous method, without the occurrence of death, Myocardial Infarction (MI), or repeat revascularization of the target lesion
Time Frame: From post-procedure up to hospital discharge
Population: Patients who were followed up to hospital discharge
Measure: Number; unit: Percentage of Participants
Arm/Group | CYPHER NxT Stent on the BX SONIC OTW SDS
Number analyzed (Participants) | 100
Percentage of Participants | 97
Statistical Analysis 1: Comparison: CYPHER NxT Stent on the BX SONIC OTW SDS; Test type: Superiority or Other; Qualitative Comparison; Reported in qualitative/semi-quantitative comparitive fashion due to study design; Percentage of participants = 97.0, 95% CI [91.5 to 99.4], Standard Error of Mean 1.71

2. Secondary Outcome: Percentage of Participants Who Experienced Any Major Adverse Cardiac Events From Post-procedure to 30 Days Later
Description: Major Adverse Cardiac Events (MACE) consists of death, Myocardial Infarction (Q-wave and Non Q-wave), emergent Coronary Artery Bypass Graft (CABG) or Target Lesion Revascularization (TLR).
Time Frame: From post-procedure up to 30 days
Population: Patients who had 30 days clinical follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | CYPHER NxT Stent on the BX SONIC OTW SDS
Number analyzed (Participants) | 99
Percentage of Participants | 3.0
Statistical Analysis 1: Comparison: CYPHER NxT Stent on the BX SONIC OTW SDS; Test type: Superiority or Other; No formal statistical testing; Percentage of participants = 3.0, 95% CI [0.6 to 8.6]

3. Secondary Outcome: Percentage of Participants Who Experienced Any Major Adverse Cardiac Events From Post-procedure to Hospital Discharge
Description: as for outcome 2
Time Frame: From post-procedure up to hospital discharge
Population: Patients who were followed up to hospital discharge
Measure: Number; unit: Percentage of participants
Arm/Group | CYPHER NxT Stent on the BX SONIC OTW SDS
Number analyzed (Participants) | 100
Percentage of participants | 3.0
Statistical Analysis 1: Comparison: CYPHER NxT Stent on the BX SONIC OTW SDS; Test type: Superiority or Other; Descriptive statistics; Percentage of participants = 3.0, 95% CI [0.6 to 8.5]

4. Secondary Outcome: Percentage of Participants Who Experienced Any Major Adverse Cardiac Events From Post-procedure to 12 Months Later
Description: as for outcome 2
Time Frame: From post-procedure up to 12 months
Population: Patients who had at least 330 days clinical follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | CYPHER NxT Stent on the BX SONIC OTW SDS
Number analyzed (Participants) | 96
Percentage of participants | 10.4
Statistical Analysis 1: Comparison: CYPHER NxT Stent on the BX SONIC OTW SDS; Test type: Superiority or Other; Descriptive statistics; Percentage of participants = 10.4, 95% CI [5.1 to 18.3]

ADVERSE EVENTS:
Arm/Group | CYPHER NxT Stent on the BX SONIC OTW SDS
Serious Adverse Events (participants affected / at risk) | 1/95
Other Adverse Events (participants affected / at risk) | 12/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYPHER NxT Stent on the BX SONIC OTW SDS (N=95)
Death (Vascular disorders) | 1 (1) — The number at risk is defined as the number of patients who had sufficient (one year) follow-up or who had an event prior to the end of follow-up.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYPHER NxT Stent on the BX SONIC OTW SDS (N=96)
Myocardial Infarction (Q wave or Non-Q wave) (Vascular disorders) | 3 (3) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.
Emergent CABG (Vascular disorders) | 1 (1) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.
Target Lesion Revascularization (Vascular disorders) | 6/95 (6) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.
Target Vessel Revascularization not involving the Target Lesion (Vascular disorders) | 1/95 (1) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.
Target Vessel Revascularization (Vascular disorders) | 7/95 (7) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.
Target Vessel Failure (Vascular disorders) | 10 (10) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.
Major Vascular Complications (Vascular disorders) | 1/95 (1) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.
Ischemic Complications (Vascular disorders) | 1 (1) — The number at risk is defined as the number of patients who had sufficient one year post-procedure follow-up or who had at least one event prior to the end of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less